CLINICAL TRIAL: NCT05233566
Title: Ketamine for Postoperative Avoidance of Depressive Symptoms: The K-PASS Feasibility Trial
Acronym: K-PASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Bradley Fritz, Instructor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202201107
Record Dates: First submitted 2022-02-03; First posted 2022-02-10 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Depression
MeSH Terms: interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Arm (Experimental): Following surgery and extubation, patients will receive ketamine 0.5 mg/kg over 10 minutes followed by an infusion of 0.3 mg/kg/h for 2 hours 50 minutes.
  Interventions: Drug: Ketamine
- Control Arm (Placebo Comparator): Following surgery and extubation, patients will receive normal saline at an equal rate to that used in the ketamine arm.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine — NMDA antagonist
  Other Names: Ketalar
  Arms: Ketamine Arm
Drug: Normal saline — IV fluid acting as a placebo
  Arms: Control Arm

SUMMARY:
This protocol describes a feasibility trial that will evaluate the feasibility of conducting a full-scale phase 3 trial testing the hypothesis that a postoperative sustained, low-dose ketamine infusion can prevent postoperative depressive symptoms when administered to a targeted population of neurosurgical patients with a history of depression.

DETAILED DESCRIPTION:
This protocol describes a feasibility trial that will evaluate the feasibility of conducting a full-scale phase 3 trial. Both the feasibility trial and the full-scale trial will follow a randomized, placebo-controlled, double-blinded, parallel design. The trial will follow a superiority design. This trial will take place at a single site (Washington University in St. Louis School of Medicine/Barnes-Jewish Hospital).

Following extubation, patients will be randomized to the intervention (ketamine group) or to control (control group). Patients in the ketamine group will receive a bolus of ketamine 0.5 mg/kg intravenously over 10 minutes, followed by an infusion at 0.3 mg/kg/h for an additional 2 hours 50 minutes. Patients in the control group will receive an equal volume of normal saline. Patients, research staff performing assessments, and research staff performing data analysis will be blinded to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written, informed consent
2. Aged 18 or older
3. Scheduled for non-ambulatory surgery scheduled to last at least 2 hours at Barnes-Jewish Hospital
4. Past medical history of depression, defined as one or more of the following criteria

   1. Previous diagnosis by a psychiatrist or primary care physician in an outpatient or inpatient setting, by patient report or chart documentation
   2. Prescription of an oral antidepressant by a psychiatrist or primary care physician for a mood disorder

Exclusion Criteria:

1. Bipolar depression
2. Concurrent use of a medication contraindicated with ketamine
3. Emergent surgery
4. Known or suspected elevation in intracranial pressure
5. Current subarachnoid hemorrhage
6. Carotid endarterectomy or arteriovenous malformation repair
7. Allergy to ketamine
8. Any condition in which a significant elevation of blood pressure would constitute a serious hazard (e.g., aortic dissection, pheochromocytoma)
9. Known history of dementia
10. Pregnancy or lactation
11. Inability to converse in English
12. Concurrent enrollment in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Fritz BA, Tellor Pennington BR, Dalton C, Horan C, Palanca BJA, Schweiger JA, Griffin L, Tumwesige W, Willie JT, Farber NB. Ketamine for postoperative avoidance of depressive symptoms: the K-PASS feasibility randomised trial. BJA Open. 2023 Dec 15;9:100245. doi: 10.1016/j.bjao.2023.100245. eCollection 2024 Mar. PMID 38179107
- [Derived] Fritz BA, Tellor Pennington BR, Palanca BJA, Schweiger JA, Willie JT, Farber NB. Protocol for the Ketamine for Postoperative Avoidance of Depressive Symptoms (K-PASS) feasibility study: A randomized clinical trial. F1000Res. 2022 May 11;11:510. doi: 10.12688/f1000research.121529.1. eCollection 2022. PMID 37483552

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine Arm | Control Arm
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Arm | Control Arm | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Full Range); unit: years] | 47.4 [23 to 75] | 48.5 [23 to 75] | 47.9 [23 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 15 | 14 | 29
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Preoperative Depressive Symptoms - Montgomery-Asberg Depression Rating Scale [Count of Participants; unit: Participants]
  0-6 (No symptoms) | 3 | 5 | 8
  7-19 (Mild symptoms) | 6 | 5 | 11
  20-34 (Moderate symptoms) | 6 | 5 | 11
  35-60 (Severe symptoms) | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Approached Patients Who Enroll and Are Randomized
Description: The numerator will include all patients who are randomized to receive either ketamine or placebo.
  The denominator will include all patients who are approached by the research team to evaluated eligibility and offer consent.
Time Frame: 3 days after surgery
Population: The analysis population for this outcome includes all patients who were approached by the research team, including those who decided not to participate in the trial and those who were excluded from the trial prior to randomization. Because these patients were never randomized, it is not possible to report results for this outcome separately for the Ketamine Arm and the Control Arm.
Measure: Count of Participants; unit: Participants
Groups:
- Protocol Version 1: Under protocol version 1, the inclusion criteria included patients aged ≥18 yr with a history of depression undergoing surgery at Barnes-Jewish Hospital with planned ICU admission.
- Protocol Version 2: Under protocol version 2, the inclusion criteria included patients aged ≥18 yr with a history of depression undergoing non-ambulatory surgery scheduled for at least 2 h.
Arm/Group | Protocol Version 1 | Protocol Version 2
Number analyzed (Participants) | 27 | 101
Participants | 1 | 31

2. Primary Outcome: Fraction of Randomized Patients Who Complete the Study Infusion
Description: The numerator will include all participants who received the entire study medication infusion as planned.
  The denominator will include all participants who are randomized to receive either ketamine or the placebo.
Time Frame: 3 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Arm | Control Arm
Number analyzed (Participants) | 16 | 16
Participants | 15 | 15

3. Primary Outcome: Fraction of Randomized Patients With Depression Rating Scale Scores at All Specified Time Points
Description: Depression will be measured using the Montgomery-Asberg Depression Rating Scale (MADRS) at pre-operative baseline and on post-infusion days 1, 2, 4, 7, and 14. MADRS scores range 0 to 60, with higher scores representing worse depression.
  The numerator will include all patients with MADRS scores documented at all 6 time points.
  The denominator will include all participants who are randomized to receive either ketamine or the placebo.
Time Frame: 14 days after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Arm | Control Arm
Number analyzed (Participants) | 16 | 16
Participants | 13 | 6

4. Secondary Outcome: Depressive Symptoms on Day 4
Description: Depression will be measured using the Montgomery-Asberg Depression Rating Scale (MADRS) at pre-operative baseline and on post-infusion days 1, 2, 4, 7, and 14. MADRS scores range 0 to 60, with higher scores representing worse depression.
  The distribution of MADRS scores in the population will be assessed for normality using visual analysis of histograms and using the Kolmogorov-Smirnoff test. If the MADRS scores are normally distributed, then the mean scores in the two groups on post-infusion day 4 will be compared using linear regression, adjusting for preoperative score. If the MADRS scores are not normally distributed, then the median delta scores in the two groups will be compared using median regression, adjusting for preoperative score.
  Participants with missing MADRS scores at either time point (preoperative baseline or post-infusion day 4) will be excluded.
Time Frame: 4 days after the intervention
Population: Excludes participants with missing MADRS scores either at baseline or on post-infusion day 4.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ketamine Arm | Control Arm
Number analyzed (Participants) | 13 | 11
score on a scale | 4 [2 to 16] | 6 [3.5 to 12]

5. Secondary Outcome: Delta Sleep Ratio on Night 1 Following Study Medication
Description: Electroencephalograms (EEG) will be captured during sleep using the Dreem headband (DREEM, Rhythm, New York, NY), a consumer-grade wireless device using dry electrodes. Sleep stages (e.g., non-rapid eye movement [NREM], rapid eye movement, wakefulness) will be detected using the Dreem headband's built-in automated sleep scoring algorithm. During each time epoch, slow wave activity will be defined as the EEG power in the range 1-4 Hz. The delta sleep ratio (DSR) will be defined as the ratio of slow wave activity during the first NREM epoch to slow wave activity during the second NREM epoch.
  Because it is a ratio, the DSR is a dimensionless number. In normal sleep, slow wave activity is greatest at the beginning of the night and decreases throughout the night. Therefore, higher DSR values reflect a more normal sleep architecture.
Time Frame: 2 days after intervention
Measure: Mean (Full Range); unit: ratio (dimensionless number)
Arm/Group | Ketamine Arm | Control Arm
Number analyzed (Participants) | 2 | 3
ratio (dimensionless number) | 3.01 [2.99 to 3.03] | 0.96 [0.20 to 1.63]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Ketamine Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/16 | 1/16
Serious Adverse Events (participants affected / at risk) | 2/16 | 5/16
Other Adverse Events (participants affected / at risk) | 0/16 | 3/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine Arm (N=16) | Control Arm (N=16)
Seizure (Nervous system disorders) | 0 | 1
Ramsay Hunt syndrome (Nervous system disorders) | 1 | 0
Postoperative Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Subjective arm/leg weakness (Nervous system disorders) | 0 | 1
Surgical Site Infection (Infections and infestations) | 0 | 1
Deep Venous Thrombosis (Blood and lymphatic system disorders) | 0 | 1
Death (underlying etiology unable to be determined) (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine Arm (N=16) | Control Arm (N=16)
Transient Ischemic Attack (Nervous system disorders) | 0 | 1
Blisters around incision (Skin and subcutaneous tissue disorders) | 0 | 1
Fever and chills (General disorders) | 0 | 1
Nausea and vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT05233566/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT05233566/ICF_001.pdf